CLINICAL TRIAL: NCT01258920
Title: A Long-Term, Open-Label Study of Flexibly Dosed Paliperidone Palmitate Long-Acting Intramuscular Injection in Japanese Patients With Schizophrenia
Brief Title: A Study of Paliperidone Palmitate in Japanese Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR017077; PALM-JPN-5 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2010-11-04; First posted 2010-12-13 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperidone palmitate; Intramascular Injection
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paliperidone palmitate (Experimental): Paliperidone palmitate Paliperidone palmitate will be administered im as an initial loading dose of 150 mg eq. on Day 1 and 100 mg eq. 1 week later in the deltoid muscle and will be administered in a flexible dose range of 25 to 150 mg eq. at 4-week intervals from Week 5 for a total of 11 injections.
  Interventions: Drug: Paliperidone palmitate

INTERVENTIONS:
Drug: Paliperidone palmitate — Paliperidone palmitate will be administered im as an initial loading dose of 150 mg eq. on Day 1 and 100 mg eq. 1 week later in the deltoid muscle, and will be administered in a flexible dose range of 25 to 150 mg eq. at 4-week intervals from Week 5 for a total of 11 injections.

SUMMARY:
The primary objective of this study is to evaluate the long-term safety and tolerability of paliperidone palmitate in Japanese patients with schizophrenia. Secondary objectives of this study are to: explore the efficacy on symptoms of schizophrenia and the maintenance of treatment effect; explore the pharmacokinetics of paliperidone palmitate through sparse pharmacokinetic sampling.

DETAILED DESCRIPTION:
This is an open-label, flexible-dose, multicenter study. The study will consist of 3 periods: an up-to-2-week pre-observation (screening) period, an observation period from Day 1 (baseline) to Week 49 (end of observation period) assessment, and a post-observation period from after the Week 49 (end-of-observation period) assessment to Week 57. For the patients who discontinue the study before the last assessment in Week 49, the post observation period will start after the discontinuation from observation period assessment with follow-up visits at 4, 8, and 12 weeks after the last injection. The total duration of the study will be 57 weeks, including the observation and post observation periods. Approximately 200 men and women, aged 20 years or older who meet the DSM-IV-TR criteria for schizophrenia at least 1 year before screening and have a Positive and Negative Syndrome Scale (PANSS) total score of 60 to 120 at screening and baseline will be enrolled, so that at least 100 patients complete this 1-year study. The patients who have a primary active Axis I disorder other than schizophrenia will not be enrolled in the study. Eligible patients will be administered an initial loading dose of paliperidone palmitate 150 mg eq. im on Day 1 and 100 mg eq. 1 week later in the deltoid muscle. The study drug will be administered in a flexible dose range of 25 to 150 mg eq. at 4-week intervals from Week 5 as either deltoid or gluteal muscle injections for a total of 11 injections. A dose of 75 mg eq. is recommended from Week 5 until Week 45. The study drug will be administered by a study drug manager and/or injector. Each dose increase should be in increments of 50 mg eq. or less. Dose increases can be considered if there is an increase in the PANSS total score (individual items or the total) or the Clinical Global Impression - Severity (CGI-S) score from the preceding assessment. Dose decreases can be considered if adverse events occur that appear to have a causal relationship with the investigational drug. The injection site (deltoid or gluteal) will, in principle, be fixed at the fourth injection and thereafter, but injection in the deltoid or gluteal muscle can be alternated at the discretion of the investigator if considered appropriate for the patient's safety. If repeated injections are administered in either the deltoid or gluteal muscles, then alternating the side of each injection (left or right) is recommended. The choice of injection needle will be determined by the patient's weight and by the injection site. The weight at baseline (Day 1) will be used when choosing needles for injection from Day 1 to Week 21, and the weight at Week 25 will be used when choosing needles for injection at Week 25 and thereafter. Patients weighing less than 200 lb (<90 kg) will receive their deltoid injection with a 1-inch needle (23 G×1"). Patients weighing 200 lb or more (=90 kg), will receive their deltoid injection with a 1.5-inch needle (22 G×1 1/2"). All gluteal injections will be administered with a 1.5-inch needle (22 G×1 1/2"). The sponsor will collect adverse events starting with the signing of the informed consent form until completion of all end-of-study procedures. Adverse events will be followed by the investigator until it recovers or is considered clinically stable. Adverse events include any occurrence that is new in onset or aggravated in severity or frequency from the baseline condition, or abnormal results of diagnostic procedures, including laboratory test abnormalities. Blood samples (preferably fasted), for serum chemistry and hematology and a random urine sample for urinalysis, electrocardiogram (ECG), vital signs, height, weight, waist circumference, Body Mass Index (BMI), Drug-Induced Extrapyramidal Symptoms Scale (DIEPSS), Columbia-Suicide Severity Rating Scale (C-SSRS), evaluation of the injection site and Visual Analog Scale (VAS) for patient's assessment of injection pain will be also collected for safety evaluation. PANSS total score and CGI-S score will be collected for efficacy evaluation. Samples for pharmacokinetic evaluation will be collected at designated timepoints. An optional 10-mL pharmacogenomic blood sample will be collected from patients who provide a separate written informed consent for this part of the study. The patients will receive paliperidone palmitate intramuscular (im) as an initial loading dose of 150 mg eq. on treatment Day 1 and 100 mg eq. 1 week later in the deltoid muscle. The study drug will be administered in a flexible dose range of 25 to 150 mg eq. at 4-week intervals from Week 5 as either deltoid or gluteal muscle injections for a total of 11 injections. A dose of 75 mg eq. is recommended from Week 5 until Week 45.

ELIGIBILITY:
Inclusion Criteria:

* Met diagnostic criteria for schizophrenia according to DSM-IV-TR (disorganized type [295.10], catatonic type [295.20], paranoid type [295.30], residual type [295.60], or undifferentiated type [295.90]) for at least 1 year before screening. Prior medical records, written documentation or verbal information obtained from previous psychiatric providers obtained by the investigator must be consistent with the diagnosis of schizophrenia
* A PANSS total score of 60 to 120 at screening and baseline (Day 1)
* Documented history of exposure to either a risperidone formulation or a paliperidone formulation and known to be tolerated before baseline (Day 1). (Even if the patient's experience of taking risperidone or paliperidone cannot be confirmed at the time of informed consent, the patient will be able to meet this criterion if the patient takes oral risperidone 2 mg/day or more or paliperidone ER 6 mg/day or more for at least 4 days between the day of informed consent and the day before baseline, and it is possible to confirm that there is no lack of tolerability in the patient)
* Women of childbearing potential must have a negative ß-human chorionic gonadotropin (ß-hCG) pregnancy test at the screening urine pregnancy test
* Patients must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

* Primary active DSM-IV-TR Axis I diagnosis other than schizophrenia
* A DSM-IV-TR diagnosis of active substance dependence within 3 months before screening (nicotine and caffeine are not exclusionary)
* Relevant history of or current presence of any significant or unstable cardiovascular, respiratory, neurological (including seizures or significant cerebrovascular), renal, hepatic, hematologic, endocrine, immunologic, or other systemic disease
* History or current presence of neuroleptic malignant syndrome or tardive dyskinesia
* Known or suspected hypersensitivity or intolerance to risperidone, paliperidone, or any of their excipients (including egg yolks, soybean oil, phospholipids, and glycerol)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2010-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events as a measure of safety and tolerability | 49 Weeks

SECONDARY OUTCOMES:
The change from baseline in Positive and Negative Syndrome Scale (PANSS) total score | Baseline, Week 49
  The PANSS is a 30-item scale designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items and ranges from 30 to 210. Higher scores indicate worsening.
The change from baseline in Clinical Global Impression - Severity (CGI-S) score | Baseline, Week 49
  The CGI-S rating scale is a 7 point global assessment that measures the clinician's impression of the severity of illness exhibited by a patient. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill patients". Higher scores indicate worsening.
Pharmacokinetic evaluations (graphically display to explore dose proportionality and achievement of steady state) | 49 Weeks (Baseline, Week 1, 5, 9, 13, 21, 25, 37, 45, 47 and 49)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (29):
- Japan (29):
  - Asahi
  - Fujioka
  - Fujisawa
  - Hachiōji
  - Higashimurayama
  - Hiroshima
  - Iizuka
  - Kanuma
  - Kashihara
  - Kashiwara
  - Kochi
  - Kure
  - Maebashi
  - Moriguchi
  - Nagasaki
  - Nirasaki
  - Ohta
  - Sapporo
  - Shimonoseki
  - Shinjyuku
  - Takatsuki
  - Tama
  - Tokushima
  - Tokyo
  - Ube
  - Ueda
  - Uji
  - Yokohama
  - Yokosuka

REFERENCES:
- See also: A Long-Term, Open-Label Study of Flexibly Dosed Paliperidone Palmitate Long-Acting Intramuscular Injection in Japanese Subjects With Schizophrenia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=437&filename=CR017077_CSR.pdf